CLINICAL TRIAL: NCT01796834
Title: Managing Diabetes Mindfully Study
Acronym: MDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23AT003919-01A2 (NIH); K23AT003919-01A2 (NIH)
Record Dates: First submitted 2013-02-19; First posted 2013-02-22 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Mindfulness-Based Stress Reduction; Diabetes Management; Stress Reduction; Diabetes Testing
MeSH Terms: conditions — Diabetes Mellitus | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mindfulness-Based Stress Reduction (Experimental): Subjects attend a community based Mindfulness-Based Stress Reduction course.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — An 8-9 week MBSR course led by an experienced instructor in a group format. Participants learn mindfulness meditation techniques and simple yoga exercises. Subjects receive four phone support calls.

SUMMARY:
To evaluate the feasibility of conducting a trial of a mindfulness-based stress reduction (MBSR) program for patients with diabetes (DM) on measures of HbA1c, blood pressure, perceived stress, depression, patient self-efficacy and quality of life; and to estimate the effect of a MBSR program for patients with DM. It is expected that MBSR program participants will evidence a trend toward better clinical outcome measures of HbA1c, blood pressure, and standardized measures of diabetes self-management, perceived stress, depression, self-efficacy, and quality-of-life.

DETAILED DESCRIPTION:
Primary Objective: Evaluate the feasibility of conducting a trial of a MBSR program for patients with diabetes on measures of HbA1c, blood pressure, perceived stress, depression, patient self-efficacy and quality of life. Feasibility will be assessed via: a) the interest of patients in taking part in an MBSR program; c) the effectiveness of strategies for recruiting patients with diabetes into the study; d) rates of participant compliance with the MBSR; and, e) patient compliance with the program evaluation plan.

Estimate the effect of a MBSR program for patients with diabetes. It is expected that MBSR program participants will evidence a trend toward better clinical outcome measures of HbA1c, blood pressure, and standardized measures of diabetes self-management, perceived stress, depression, self-efficacy, and quality-of-life.

Secondary Objective: To explore the experience of people with diabetes who participate in an MBSR course through the use of semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* English speaking
* have type 2 diabetes, with 2 HbA1C values >8 in prior 16 months
* HbA1C value of >8 within 3 months of intervention start
* able to read course materials
* mentally intact with no history of mental illness or major depression
* reachable by phone (for phone support component)
* able to attend weekly classes
* willing to provide written informed consent

Exclusion Criteria:

* completed formal training in other mind body practices such as meditation, yoga, or tai chi within the prior year or currently have a regular ongoing practice in this area.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
HbA1C Blood Test | Baseline and 12-15 weeks from start of intervention period
  This HbA1C blood test will be compared to a qualifying HbA1C blood test.

SECONDARY OUTCOMES:
Blood Pressure | 8 weeks during intervention
  Subjects will self-administer blood pressure testing with a wrist blood pressure cuff and a Daily Log provided to the subject and record results during the intervention period.

OTHER OUTCOMES:
Measures of diabetes self-management | At baseline and 0 - 3 weeks after completion of the intervention
  By self report (survey)
Measure of perceived stress | At baseline and 0 - 3 weeks after completion of the intervention
  By self report (survey)
Measure of depression | At baseline and 0 - 3 weeks after completion of the intervention
  By self report (survey)
Measure of self-efficacy | At baseline and 0 - 3 weeks after completion of the intervention
  By self report (survey)
Measure of quality of life | At baseline and 0 - 3 weeks after completion of the intervention
  By self report (survey)
patient evaluation of MBSR intervention | week 12- 15 post baseline measures
  semi-structured telephone interviews with subjects evaluating their perception of the value of the intervention on their overall diabetes management; their satisfaction with the intervention; and their perception of the intervention impact on their quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Robin Whitebird, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Institute for Education and Research, Bloomington, Minnesota, United States

REFERENCES:
- [Derived] Whitebird RR, Kreitzer MJ, Vazquez-Benitez G, Enstad CJ. Reducing diabetes distress and improving self-management with mindfulness. Soc Work Health Care. 2018 Jan;57(1):48-65. doi: 10.1080/00981389.2017.1388898. Epub 2017 Oct 24. PMID 29064772